CLINICAL TRIAL: NCT04310813
Title: Microscopic-spectroscopic Examination for Urothelial Tissue Characterization
Acronym: MSUT
Status: Completed | Type: Observational
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, Gianluca Villa, MD, clinical researcher, Careggi Hospital
Other Study IDs: CEAVC 10325/2016
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Bladder Tumor
Keywords: Bladdder Cancer; Urothelial tumor; Pathology; Spectroscopy; BCa
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic urologic patients: Patients with bladder cancer or benign prostate hyperplasia undergoing urologic endoscopic procedures.
  Interventions: Diagnostic Test: Multimodal spectroscopic analysis

INTERVENTIONS:
Diagnostic Test: Multimodal spectroscopic analysis — During time of bladder or prostate resection, freshly excised cold cup biopsies of both bladder cancer or healthy bladder mucosa were taken and sent for inspection through label-free multimodal fiber optic spectroscopy (MFOS) within 30 minutes

SUMMARY:
To evaluate the possibility to properly discriminate between healthy bladder tissue and BCa with a multimodal fiber optic spectroscopy (MFOS) technique, in order to possibly introduce a more objective way to detect BCa, thus reducing inter-observer variability and maybe to determine urothelial carcinoma stage and grade with a comparable accuracy, specificity and sensibility of the current gold standard histopathological analysis

DETAILED DESCRIPTION:
Observational single center study on human biological samples to evaluate the possibility to discriminate between healthy and tumor tissue on urothelial bladder samples. Aim of the study is to provide a fast, reliable and label free aid/alternative to current histopathology

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate,
* legal age,
* full capacity to sign informed consent
* eligibility for each surgical operation according to the best clinical practice and the urological guidelines

Exclusion Criteria:

* concomitant use of Hexaminolevulinate (Hexvix®)
* concomitant ongoing UTIs,
* concomitant bladder stone presence,
* recent catheterization or persistent bladder catheterization at time of surgery,
* concomitant presence of other pelvic cancer (both prostate, urethral, uterine),
* previous chemotherapy or radiotherapy of the pelvis,
* patient refusal at informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled at hospitalization in our Urology Ward for surgical operation. Patients in surgical note for TURBT for bladder cancer or for Trans-Urethral Resection of Prostate (TURP) for Benign Prostatic Hyperplasia (BPH) are prospectively enrolled.
  Age, history of bladder cancer, smoke habit and anamnesis are recorded before surgery. During time of bladder or prostate resection, freshly excised cold cup biopsies of both bladder cancer or healthy bladder mucosa are taken and sent for inspection through label-free multimodal fiber optic spectroscopy (MFOS) within 30 minutes.
  Specimens are sent to standard histopathological analysis. MFOS data are then compared to current gold standard methodology in order to develop a classification algorithm based on the spectral information provided by each technique.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
diagnostic concordance | 30 minutes from resection
  concordance in identifying healthy and tumor tissue between multimodal fiberoptic spectroscopy and pathology, considered as gold standard

SECONDARY OUTCOMES:
grading concordance | 30 minutes from resection
  concordance in discriminating low vs high grade tumor between multimodal fiberoptic spectroscopy and pathology, considered as gold standard
staging concordance | 30 minutes from resection
  concordance in discriminating Ta vs T1 vs T2 tumors between multimodal fiberoptic spectroscopy and pathology, considered as gold standard

CONTACTS AND LOCATIONS:
Overall Officials: Simone Morselli, MD, Study Chair — University of Florence

IPD SHARING:
Plan to Share IPD: No